CLINICAL TRIAL: NCT06433674
Title: Enteral Zinc Supplementation in Very Low Birth Weight Infants
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-09580-FB
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Very Low Birth Weight Infant; Nutritional Deficiency
MeSH Terms: conditions — Malnutrition | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: The intervention will be two parallel groups. one Group receiving Zinc Sulfate. The other group receiving Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zinc Sulfate (Experimental): The experimental group will receive ~1 mg/kg/day of elemental enteral Zinc
  Interventions: Drug: Zinc Sulfate
- Placebo (Placebo Comparator): The placebo group will receive a similar amount of sterile water in a colored syringe
  Interventions: Other: Sterile Water

INTERVENTIONS:
Drug: Zinc Sulfate — The pharmacy will be the one preparing the Zinc sulfate. The zinc sulfate comes in 220 mg tablets which are then mixed with 1 ml of Oral plus (a common suspending agent) as well as 9 ml of Sterile water. This then makes a Zinc Sulfate 22 mg/ml oral suspension which will be dispensed in an amber syringe.
  Arms: Zinc Sulfate
Other: Sterile Water — The placebo group with will receive a similar amount of sterile water in a colored syringe
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to observe for changes in rate of weight gain in the very low birth weight (VLBW) infants by adding an enteral Zinc supplement of 1 mg/kg/day of elemental zinc. The main question it aims to answer:

• Does an enteral Zinc supplement of 1 mg/kg/day increase rate of weight gain in VLBW infants Researches will compare the experimental group to a placebo group to see if there is a statistical difference in rate of weight gain between the two groups

* Once the participants have reached 100 ml/kg/day of enteral feeds. The participants will be randomized to one of two groups. The treatment group will receive ~1 mg/kg/day of elemental enteral Zinc, and the control group to receive similar amount of enteral sterile water put in a colored syringe. The Zinc Supplement would be Zinc Sulfate. The primary team would otherwise be managing the patient's feeding using our hospital's feeding protocol. As long as the patient is tolerating 100 ml/kg/day of enteral feeds, the Zinc Supplement will continue until 36 weeks postmenstrual age (PMA) or hospital discharge, whichever comes first.
* The participants will have three Zinc levels measured: once prior to Zinc Supplementation, once at around the four week mark, and once at the completion of therapy.

DETAILED DESCRIPTION:
This is a prospective, single center, randomized, double blinded, placebo controlled clinical trial. The goal of this clinical trial is to observe for changes in rate of weight gain in the VLBW infants by adding an enteral Zinc supplement of 1 mg/kg/day of elemental zinc. The main question it aims to answer:

• Does an enteral Zinc supplement of 1 mg/kg/day increase rate of weight gain in VLBW infants Researches will compare the experimental group to a placebo group to see if there is a statistical difference in rate of weight gain between the two groups

* Once the participants have reached 100 ml/kg/day of enteral feeds. The participants will be randomized using sealed envelopes. The subjects will be randomly selected to one of two groups. The treatment group will receive ~1 mg/kg/day of elemental enteral Zinc, and the control group to receive similar amount of enteral sterile water put in a colored syringe. The Zinc Supplement would be Zinc Sulfate. Only the pharmacy will know which patient is receiving the Zinc Sulfate and which patient is receiving the placebo. The primary team would otherwise be managing the patient's feeding using our hospital's feeding protocol. As long as the patient is tolerating 100 ml/kg/day of enteral feeds, the Zinc Supplement will continue until 36 weeks PMA or hospital discharge, whichever comes first.
* The participants will have three Zinc levels measured: once prior to Zinc Supplementation, once at around the four week mark, and once at the completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight < 1500 grams
2. Infant is tolerating at least 100 ml/kg/day of enteral feeds
3. At least 25wks PMA.

Exclusion Criteria:

* Major congenital malformations especially anomaly of the GI tract
* Major congenital heart disease (i.e.: ductal dependent lesion)
* Previously diagnosed necrotizing enterocolitis (stage 2 or 3), bowel perforation, or bowel resection
* Infant who has tolerated ≥100 ml/kg/day prior to admission.

Ages: 25 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of weight gain | at hospital discharge or 36 weeks PMA whichever comes first.
  The primary outcome would be the rate of weight gain in grams/kg/day

SECONDARY OUTCOMES:
Length | at hospital discharge of 36 weeks PMA whichever comes first
  This secondary outcome would be the rate of length gain in cm/day
Head Circumference | at hospital discharge of 36 weeks PMA whichever comes first
  This secondary outcome would be the rate of head circumference gain in cm/day
Zinc level | Comparing the initial zinc level to the four week zinc level as well as the zinc level at 36 weeks or discharge whichever comes first
  This secondary outcome would be looking for a statically significant difference in zinc level

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Mire, M.D., Principal Investigator — UTHSC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terrin G, Berni Canani R, Passariello A, Messina F, Conti MG, Caoci S, Smaldore A, Bertino E, De Curtis M. Zinc supplementation reduces morbidity and mortality in very-low-birth-weight preterm neonates: a hospital-based randomized, placebo-controlled trial in an industrialized country. Am J Clin Nutr. 2013 Dec;98(6):1468-74. doi: 10.3945/ajcn.112.054478. Epub 2013 Sep 11. PMID 24025633
- [Background] Brion LP, Heyne R, Lair CS. Role of zinc in neonatal growth and brain growth: review and scoping review. Pediatr Res. 2021 May;89(7):1627-1640. doi: 10.1038/s41390-020-01181-z. Epub 2020 Oct 3. PMID 33010794
- [Background] Terrin G, Berni Canani R, Di Chiara M, Pietravalle A, Aleandri V, Conte F, De Curtis M. Zinc in Early Life: A Key Element in the Fetus and Preterm Neonate. Nutrients. 2015 Dec 11;7(12):10427-46. doi: 10.3390/nu7125542. PMID 26690476
- [Background] Sinha B, Dudeja N, Chowdhury R, Choudhary TS, Upadhyay RP, Rongsen-Chandola T, Mazumder S, Taneja S, Bhandari N. Enteral Zinc Supplementation in Preterm or Low Birth Weight Infants: A Systematic Review and Meta-analysis. Pediatrics. 2022 Aug 1;150(Suppl 1):e2022057092J. doi: 10.1542/peds.2022-057092J. PMID 35921675
- [Result] Shaikhkhalil AK, Curtiss J, Puthoff TD, Valentine CJ. Enteral zinc supplementation and growth in extremely-low-birth-weight infants with chronic lung disease. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):183-7. doi: 10.1097/MPG.0000000000000145. PMID 24121149